CLINICAL TRIAL: NCT01054365
Title: Same Day Discharge After Coronary Stenting Trial
Status: Completed | Type: Observational
Sponsor: Leonardo Clavijo (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Leonardo Clavijo, Director of Interventional Cardiology, University of Southern California
Organization: University of Southern California (Other)
Other Study IDs: Rev 09-20-09
Record Dates: First submitted 2010-01-19; First posted 2010-01-22 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2010-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Delayed Discharge Group (DDG): D/C at least 24 hours after procedure or at usual discharge time (n =200)
- Early Discharge Group (EDG): D/C 6 hours after procedure if no indication for extended stay after randomization (n=200)

SUMMARY:
In comparison to delayed hospital discharge, a strategy of early hospital discharge of patients who undergo single and multivessel stenting for type A, B, and C lesion(s) using thienopyridine and a hemostatic femoral closure device, is associated with similar clinical outcomes, but greater patient satisfaction and similar cost.

DETAILED DESCRIPTION:
This study will be a single center prospective, randomized, non-inferiority study of four-hundred patients with stable and unstable angina (CCS class I-IV), type A, B, C lesion(s), single and multivessel disease undergoing single or multivessel coronary artery stenting. All patients will be screened and consented prior to the coronary artery stenting procedure. All patients will receive an oral bolus of a thienopyridine as pre-treatment or immediately after stent implantation. All patients will be anticoagulated with bilvalirudin or heparin during the procedure. Common femoral angiography will be performed at the end of the procedure via the side-arm of the sheath in the ipsilateral oblique view (20-40°). In patients with visible atherosclerotic disease or small common femoral arteries on angiography the size and/or the degree of stenosis will be measured by quantitative angiography. Hemostasis of the femoral-arteriotomy access site will be facilitated by deployment of a hemostatic closure device (StarClose or ProGlide). Patients will be screened and consented prior to cardiac catheterization. If the stenting procedure is performed without complications and the hemostatic closure device successfully deployed the patient will then be evaluated four hours after the completion of the procedure; if there are no complications and the patient is able to ambulate, he/she will be randomized and enrolled into either the early discharge group (EDG) or the delayed discharge group (DDG). Subjects will not be considered enrolled into the study until they have been successfully randomized into either the EDG or DDG group. Patients in the early discharge group (EDG, n=200) will be dismissed from the hospital six hours after hemostatic closure device deployment if the vital signs are stable, no bleeding complications are present, are ambulatory, there are no electrocardiographic changes suggestive of myocardial ischemia and/or arrhythmia and are free of chest pain. Patients in the delayed discharge group (DDG, n=200) will be dismissed from the hospital after the procedure at the discretion of the attending cardiologist but no sooner than 24 hours after PCI. Patients with an indication for extended hospital stay will not be discharged regardless of randomization. A detailed screening log will be kept to track the number of patients screened and consented and will include reason for screening failure (exclusion criteria, procedure related complications, closure device failure, access complication, chest pain, arrhythmias, hemodynamic instability, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing single and multivessel stenting of type A, B, and C de novo lesion(s) for the treatment of stable and unstable angina (CCS class I-IV).
* Patients will be treated with thienopyridine oral bolus, either as a pre-treatment or immediately after stenting, and recommended to be continued on daily.
* Patients will be anticoagulated with intravenous heparin or bilvalirudin during the procedure and stopped immediately after completion of the procedure.

Arterial access via the femoral artery (Sheath 5, 6, 7 or 8 French) and an arteriotomy site suitable for hemostatic device closure. Suitability for closure, defined as at least 5 mm from a bifurcation, puncture must not include the artery femoralis profunda or the superficial femoral artery, TIMI III coronary flow upon completion of the intervention and Left ventricular ejection fraction (LVEF) less than 40 per cent.

* Patients who live less than an hour away from the hospital.

Exclusion Criteria:

* Age less than 30 years old or greater than 80 years old
* Acute STEMI
* Non-STEMI with documented troponin greater than 10 at presentation to the catheterization laboratory
* Cardiogenic shock or hemodynamic instability
* Severe valvular heart disease
* Any contraindication to anticoagulation
* Pregnancy
* Patients with bleeding diathesis (including thrombocytopenia (platelets less than 100,000), thrombasthenia, Von WilleBrand's disease, or anemia (Hgb less than 10 mg per dl, Hct less than 30) or coagulopathy
* Patients with a Creatinine greater than 1.5 mg/ml
* Patients with an INR greater than 1.5
* Patients with cancer or autoimmune disease
* Patients who live greater than 60 minutes away from the hospital
* Patients who will not be able to follow-up
* Patients with inadequate social or home support (homeless, lives alone, etc)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include four-hundred consented patients undergoing percutaneous coronary stenting at the University of Southern California Hospital or LA County Hospital, patients in the study group will be discharged the day of the procedure whereas patients in the control group will be discharged at the discretion of the attending cardiologist not earlier than 24 hours after their procedure. Patients will be stratified on the basis of their initial clinical presentation, as determined by the medical history, physical examination, ECG and laboratory studies. Patients must be hemodynamically stable, and able to understand and sign an informed consent.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To compare the strategies, outcomes, and complication rates of early (same day) vs. delayed (day after the procedure) hospital discharge in patients undergoing single and multivessel stenting of type A, B, and C lesions. | Patients will be followed through hospital course, at 24-72 hours, 7-14 days post discharge and at 30-45 days for clinical evaluation via telephone contact or office visit.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Clavijo, MD, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States